CLINICAL TRIAL: NCT02840409
Title: A Phase II, Open-Labeled, Multi-Center, Randomized Controlled Trial of Vinblastine +/- Bevacizumab for the Treatment of Chemotherapy-Naïve Children With Unresectable or Progressive Low Grade Glioma (LGG)
Brief Title: Vinblastine +/- Bevacizumab in Children With Unresectable or Progressive Low Grade Glioma (LGG)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Principal Investigator, Eric Bouffet, Staff Physician, Paediatric Neuro-Oncology Program, The Hospital for Sick Children
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1000052116
Record Dates: First submitted 2016-01-28; First posted 2016-07-21 (Estimated); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Low Grade Glioma
MeSH Terms: interventions — Vinblastine; Bevacizumab

STUDY DESIGN:
Intervention Model Description: Cross over to bevacizumab-vinblastine allowed in case of progression on vinblastine only
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Active Comparator): 68 weeks of single agent Vinblastine administered once weekly IV
  Interventions: Drug: Vinblastine
- Arm B (Experimental): 68 weeks of Vinblastine administered weekly IV with the addition of 12 doses of Bevacizumab administered every two weeks IV for the initial 24 weeks.
  Interventions: Drug: Vinblastine; Drug: Bevacizumab

INTERVENTIONS:
Drug: Vinblastine
Drug: Bevacizumab
  Other Names: Avastin
  Arms: Arm B

SUMMARY:
This is an open-label, randomized, multi-center, comparator Phase II trial looking at the addition of Bevacizumab to Vinblastine in chemotherapy naïve pediatric patients with progressive Low Grade Glioma aged 6 months to less than18 years of age at the time of initiation of therapy. Participants will be randomized to Arm A or Arm B. Arm A includes 68 weeks of single agent Vinblastine administered once weekly IV. Arm B includes 68 weeks of Vinblastine administered weekly IV with the addition of 12 doses of Bevacizumab administered every two weeks IV for the initial 24 weeks. Randomization will take place at the time of registration taking into account NF1 and BRAF-KIAA1549-fusion status.

ELIGIBILITY:
Inclusion Criteria:

1. Children and adolescents aged 6 months to < 18 years old with Low Grade Glioma (See Appendix I).
2. All patients must submit tumour tissue (fresh tumour tissue is recommended) and have pathological confirmation of LGG and determination of BRAF characteristics from the Hospital for Sick Children. Exceptions will be made for patients with neurofibromatosis type 1 who have not previously had a biopsy. NF1 patients are eligible without tissue confirmation but must have definitive clinical or radiographic evidence of tumour progression or risk for significant neurologic deterioration requiring immediate therapy. If a tissue sample for NF1 patients is available from a previous biopsy, it is required to be submitted for Central Review at the Hospital for Sick Children. Please refer to the lab manual for further details.
3. Patients must have progressive disease following surgical excision based on clear radiological or clinical evidence of progression, or an incomplete excision (< 95% or > 1.0 cm2 residual tumour) with necessity to begin treatment because of a risk of neurological impairment with progression.
4. All patients on study must have measurable tumour (>1.0 cm2 of residual tissue if resection has been performed) within 28 days of enrollment.
5. Patients must have received no prior therapy including chemotherapy, biological modifiers and/or radiation treatment for the tumour with the exception of surgery.
6. Patient is able to start treatment within 14 working days after randomization.
7. Post pubertal teenagers who are sexually active agree to use two methods of contraception during the treatment period and for at least 6 months after the last dose of study drug. Please refer to Appendix V for a list of acceptable methods of contraception.
8. Lansky performance status > 50% for patients < 16 years of age. Karnofsky performance status > 50% for patients ≥ 16 years of age.
9. Patients with neurologic deficits must have deficits that are stable for a minimum of 1 week prior to enrollment.
10. Patients receiving corticosteroids must be on a stable or decreasing dose for at least 1 week prior to enrollment.
11. Life expectancy > 2 months at the time of enrollment.
12. Parents/guardians must provide written informed consent and to agree that they (and the patient) will comply with the study protocol.
13. Written assent by patient according to institutional guidelines.
14. Patients must have adequate bone marrow function within 2 weeks prior to enrollment:

    * Hemoglobin ≥ 10 g/dL (may be supported )
    * Neutrophil count ≥ 1.0 × 109/L
    * Platelet count ≥ 100 × 109/L (transfusion independent)
15. Patients not on a therapeutic dose of an anti-coagulant must have an INR ≤ 1.5 and an aPTT ≤ 1.5x institutional ULN for age within 2 weeks prior to enrollment. Anti-coagulation is permitted prior to enrollment on the condition that the patient is, according to the local clinical practice guidelines or approved product labeling, adequately anti-coagulated prior to enrollment.
16. Patients must have satisfactory liver function within 2 weeks prior to enrollment:

    * AST ≤ 3x institutional ULN for age
    * ALT ≤ 3x institutional ULN for age
    * Total Bilirubin ≤ 1.5x institutional ULN for age
17. Patients must have satisfactory renal parameters and meet the following criteria within 2 weeks prior to enrollment :

    * Serum creatinine must be ≤ 1.5x ULN for age. If the serum creatinine is > 1.5 × ULN, the glomerular filtration rate (either estimated or formal) must be >90 mL/min/1.73 m2, for patient to be enrolled.
    * Absence of clinically significant proteinuria, as defined by screening of the early morning urine (urine protein < 1g/L and/or albumin/creatinine ratio < 1.0 (mg/mmol)). If urine protein ≥ 1g/L, then Urine Protein Creatinine (UPC) ratio should be calculated. If UPC ratio > 0.5, 24-hour urine protein should be obtained and the level should be < 1000 mg/24 hours for patient enrollment. Note: UPC ratio of spot urine is an estimation of the 24 urine protein excretion - a UPC ratio of 1 is roughly equivalent to a 24-hour urine protein of 1 g. UPC ratio is calculated using one of the following formulas:

[urine protein]/[urine creatinine] - if both protein and creatinine are reported in mg/dL or [(urine protein) x0.088]/[urine creatinine] - if urine creatinine is reported in mmol/L

Quality of Life Correlative Study Inclusion Criteria (Optional):

1. Age ≥ 3 and < 18 years.
2. English- or Spanish-speaking.
3. No known history of a significant neurodevelopmental disorder prior to diagnosis of LGG (e.g., Down syndrome, Fragile X, William's Syndrome, mental retardation). Patients with NF1 are not excluded.
4. No significant motor or sensory impairment that would prevent computer use and perception of the visual and auditory test stimuli.

Exclusion Criteria:

1. Children under 6 months of age.
2. Pregnant or lactating females.
3. Use of any investigational agent, systemic, targeted or immunotherapy prior to the first dose of study treatment.
4. Any bleeding diathesis or significant coagulopathy at risk of bleeding (i.e. in the absence of therapeutic anticoagulation).
5. Patients with evidence of new symptomatic CNS hemorrhage (> grade I) on baseline MRI.
6. Any significant cardiovascular disease, e.g. aortic aneurysm requiring surgical repair or recent arterial thrombosis, CVAs, transient ischemic attacks (TIAs), and systemic hypertension (i.e., a systolic and diastolic BP ≥ 95th percentile for age, sex), prior history of hypertensive crisis or hypertensive encephalopathy or stroke, uncontrolled cardiac arrhythmia within 6 months prior to enrollment .
7. Any previous venous thromboembolism Grade 3 or higher (NCI CTCAE v. 4.03).
8. History of abdominal fistula, GI perforation, intra-abdominal abscess or active GI bleeding within 6 months prior to the first study treatment.
9. Unresolved infection.
10. An active peptic or duodenal ulcer.
11. Major surgical procedure (see Table 3 section 6.1.7), brain surgery, open biopsy or significant traumatic injury within 28 days prior to enrollment or the anticipation of the need for major (elective) surgery during the course of the study treatment.
12. Intermediate surgical procedure (see Table 3 section 6.1.7) within 2 weeks of enrollment.
13. Minor surgical procedures (see Table 3 section 6.1.7) within 3 days prior to the start of treatment (including the placement of a central line, including PICC line). Insertion of a port-a-cath will require a 7-day interval prior to the start of treatment.
14. Non-healing surgical wound.
15. A bone fracture that has not satisfactorily healed.
16. Concomitant use of the following:

    * Aspirin (> 325mg/day) within 10 days of enrollment
    * Clopidogrel (> 75mg/day) within 10 days of enrollment
    * Use of therapeutic oral or parenteral anticoagulants or thrombolytic agents for therapeutic purposes with INR and aPTT outside therapeutic standards according to institutional guidelines within 10 days of first dose of Bevacizumab. Note: The use of full-dose oral or parenteral anticoagulants is permitted as long as the INR or aPTT is within therapeutic limits (according to the medical standard of the institution) and the patient has been on a stable dose of anticoagulants for at least two weeks at the time of the Baseline Visit. Prophylactic use of anticoagulants is allowed.
17. Hypersensitivity to Chinese hamster ovary (CHO) cell products or other recombinant human or humanized antibodies.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 109 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the addition of Bevacizumab to Vinblastine compared with Vinblastine alone in chemotherapy-naïve pediatric patients with unresectable or progressive Low Grade Gliomas as measured by Response Rate (RR). | 6 months from randomization
  Objective response rate within 6 months of randomisation

SECONDARY OUTCOMES:
Overall survival (OS) at the end of study. | From the date of study completion (approximately 6.5 years (78 months)) up till the date of death.
  overal survival at 5 years post randomisation
To determine 6 month, 12 month and 2 year progression free survival (PFS) between vinblastine alone versus in combination with Bevacizumab. | At 6 and 12 months and 2 years
  Optical Coherence Tomography (OCT) should occur in conjunction with the Visual Field/Acuity exams for participating institutions equipped with OCT.
To evaluate the difference in visual outcome measures in children with optic pathway gliomas treated with vinblastine alone or in combination with Bevacizumab. | Every 3 months during treatment, every 3 months for 1 year after completion of treatment, then every 6 months for 4 years.
  visual acuity measure with Teller Grading Acuity
To determine if the prevalence of cognitive deficits in children and adolescents treated for LGG, is significantly higher than the normative population (> 14%) using the NIH Toolbox Cognitive Battery. | At 1 year off therapy
  Domains include: working memory, executive function, processing speed, episodic memory, and attention
To determine the effects of Bevacizumab on cognitive function in the pediatric population using the NIH Toolbox Cognitive Battery. | During treatment, 28 days after completing treatment, at 6 months and 1 year off therapy
  The effects of Bevacizumab on cognitive function in the pediatric
To determine if the prevalence of QOL difficulties in children and adolescents treated for LGG at 1 year off therapy, is significantly higher than the normative population (> 14%). | At 1 year off therapy
  Domains include: fatigue, physical activity, anxiety, depression, and peer relationships.

OTHER OUTCOMES:
To evaluate the safety of the combination of Vinblastine and Bevacizumab compared with Vinblastine alone in pediatric patients with LGG, focusing on serious adverse events as assessed by CTCAE v 4.03. | Through study completion which is approximately 6.5 years (78 months)
  Collection of Adverse events in the bevacizumab arm
To define and describe the toxicities of the agents in combination and of single agent Vinblastine in this treatment naïve population as assessed by CTCAE v 4.03. | Through study completion which is approximately 6.5 years (78 months)
  Collection of Adverse events in the vinblastine arm
To evaluate the effect of Bevacizumab on growth and puberty by recording patient's height and using the Tanner Scale to measure puberty. | Baseline, 28 days off therapy, and then annually for 5 years off therapy
  Growth will be analyzed by recording patient's height, following treatment until completion of puberty. Puberty will be measured using the Tanner Scale where Tanner stage V for pubic hair, breast, and genitalia represent mature development and completion of puberty.
To evaluate the effect of Bevacizumab on fertility. This includes the risk of delay in pubertal development as well as abnormal menstrual status and the risk of primary or secondary amenorrhea and later on the potential effect on pregnancies) assessed by | Baseline, 28 days off therapy, and then annually for 5 years off therapy
  Follow-up of patients regardign fertility
To prospectively determine the role of BRAF mutation/fusion in PLGG and correlate this with outcome and response to therapy. | Tissue will be submitted prior to study registration for pathology review.
  Evaluation fo response according to molecular status of the tumour
To determine the presence and prognostic significance of other mutations, including RAF1, FGFR1, MYB, MYBL1, PTPN11, NTRK2, H3F3A, ATRX and CDNK2A deletions among others. | Blood samples will be collected at Baseline.
  Evaluation fo biomarkers in the blood
To stratify PLGG based on methylation profile, using methylation arrays. | Through study completion which is approximately 6.5 years (78 months)
  Analysis of methylation profile
To determine demographic (e.g., SES, gender), disease (e.g., risk status), treatment, and behavioral predictors of neurocognitive and QOL deficits as measured by the NIH Toolbox Cognitive and PROMIS batteries in children and adolescents with LGG. | Through study completion which is approximately 6.5 years (78 months)
  Evaluation of cognitive impact of treatment
To determine the prevalence of cognitive deficits in PLGG population. | Through study completion which is approximately 6.5 years (78 months)
  Evaluation of cognitive impact of tumour and treatment
To examine the role of vascularity (including MVD) in PLGG and investigate potential biomarkers to assist in determining the population of best responders to anti-angiogenic therapy in PLGG. | Through study completion which is approximately 6.5 years (78 months)
  Analysis of biomarkers of angiogenesis
To assess the use of novel MR biomarkers to assess disease response in these patients and to correlate these with traditional imaging tools. | Through study completion which is approximately 6.5 years (78 months)
  Evaluation of MRI biomarkers of response

CONTACTS AND LOCATIONS:
Overall Officials: Eric Bouffet, MD, Principal Investigator — The Hospital for Sick Children
Locations (21):
- United States (5):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- Australia (5):
  - Children's Hospital at Westmead, Westmead, New South Wales
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Women's and Children's Hospital, North Adelaide, South Australia
  - Royal Children's Hospital, Parkville, Victoria
  - Perth Children's Hospital, Nedlands, Western Australia
- Canada (10):
  - Alberta Children's Hospital, Calgary, Alberta
  - Stollery Children's Hospital, Edmonton, Alberta
  - BC Children's Hospital, Vancouver, British Columbia
  - Cancer Care Manitoba, Winnipeg, Manitoba
  - McMaster Children's Hospital, Hamilton, Ontario
  - Children's Hospital - London Health Sciences Centre, London, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Montreal Children's Hospital, Montreal, Quebec
  - CHU du Quebec-Universite Laval, Québec, Quebec
- Starship Children's Hospital, Grafton, Auckland, New Zealand